CLINICAL TRIAL: NCT06105528
Title: A Phase 1a, Double-Blind, Placebo-Controlled, Single Ascending Dose Study of the Safety, Tolerability and Pharmacokinetics of PMN310 Infusions in Healthy Volunteers
Brief Title: A Phase 1a Study of PMN310 In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ProMis Neurosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: PMN310-101
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Results first posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Healthy Participants

STUDY DESIGN:
Intervention Model Description: There will be 5 sequential escalating dose cohort groups. Dose groups are 175 mg, 350 mg, 700 mg, 1400 mg and 2800 mg (optional) administered as a single 60-minute infusion.
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 PMN310 175mg or placebo (Experimental): PMN310 175mg or placebo administered as a 60-minute infusion.
  Interventions: Drug: PMN310; Drug: Placebo
- Cohort 2 PMN310 350mg or placebo (Experimental): PMN310 350mg or placebo administered as a 60-minute infusion.
  Interventions: Drug: PMN310; Drug: Placebo
- Cohort 3 PMN310 700mg or placebo (Experimental): PMN310 700mg or placebo administered as a 60-minute infusion.
  Interventions: Drug: PMN310; Drug: Placebo
- Cohort 4 PMN310 1400mg or placebo (Experimental): PMN310 1400mg or placebo administered as a 60-minute infusion.
  Interventions: Drug: PMN310; Drug: Placebo
- Cohort 5 PMN310 2800mg or placebo (Experimental): PMN310 2800mg or placebo administered as a 60-minute infusion.
  Interventions: Drug: PMN310; Drug: Placebo

INTERVENTIONS:
Drug: PMN310 — 60-minute intravenous infusion
Drug: Placebo — 60-minute intravenous infusion

SUMMARY:
This first in human Phase 1a clinical trial will evaluate the safety, tolerability, and pharmacokinetics of a single IV infusion of PMN310 in healthy volunteers.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled study will evaluate the safety, tolerability and pharmacokinetics of single ascending doses of intravenous PMN310 in healthy adult volunteers.

Subjects will be randomly assigned to receive either a single infusion of PMN310 or placebo. After randomization on Day 1, study drug will be administered followed by the collection of safety, tolerability, and PK data.

All dose cohorts will have lumbar punctures (LPs) for PK analysis performed on Day 3 and Day 29. Primary PK and CSF data will be obtained from Day 1 to Day 29. Safety and tolerability will be collected at all visits. The study is an 85-day study with one optional follow up assessment at Day 120.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects of childbearing potential must not be breastfeeding and must have no plans to become pregnant during the course of the study through 120 days after infusion of study drug.
2. Female subjects of non-childbearing potential must have evidence from their medical history indicating that they are not of childbearing potential.
3. Any non-vasectomized male subjects must agree to use barrier contraceptives (male or female partner condom, diaphragm, cervical cap, sponges) plus spermicide.
4. Medically healthy with no clinically significant or relevant abnormalities in medical history, physical exam, vital signs, ECG, or laboratory evaluations.
5. Has provided written informed consent.
6. Body mass index is between 18 and 32 kg/m2 (inclusive).
7. Screening MRI normal.

Exclusion Criteria:

1. Clinically significant 12-lead ECG abnormality at Screening.
2. Systolic blood pressure > 150 bpm or diastolic blood pressure > 90 bpm at Screening.
3. Experienced a significant systemic illness within 30 days of the first dose of study drug.
4. Current or relevant history of physical or psychiatric illness, any medical disorder that may require treatment or make the subject unlikely to fully complete the study, or any condition that presents undue risk from the investigational product or procedures.
5. Currently using any medication except for acetaminophen as needed for miscellaneous aches and pains.
6. History of alcohol abuse and/or illicit drug use within 12 months prior dosing or a smoking history (use of tobacco products).
7. Unwilling to refrain from ingesting alcohol within the limits required by the Study.
8. Positive urine drug screen.
9. History of prior malignancy.
10. Documented history of human immunodeficiency virus (HIV) antibody or tested positive for hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibody at Screening.
11. Donated blood or blood products (e.g., plasma, platelets) within 28 days prior to first dose.
12. Received an investigational agent within the last 30 days or 5 half-lives (if known) prior to Screening, whichever is longer.
13. Contraindication to brain venipuncture, MRI or LP.
14. Indication of potential suicidality risk as identified by the following Columbia-Suicide Severity Rating Scale (C SSRS).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-11-18 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Fernandez, MD, Principal Investigator — Clnical Pharmacology of Miami; Alexander N Prezioso, MD, Principal Investigator — Clnical Pharmacology of Miami; Angela Eakin, MD, Principal Investigator — Ohio Clinical Trials
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - Ohio Clinical Trials, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: To evaluate the short-term safety and tolerability of PMN310, each cohort enrolled a sentinel group of 2 subjects who were dosed prior to dosing the remaining 6 subjects in the cohort (5:1, PMN310:placebo).A total of 129 subjects were screened, of whom, 40 subjects were randomized to treatment groups as follows: 6 subjects each in the PMN310 175 mg, 350 mg, 700 mg, 1400 mg, and 2800 mg groups and 2 subjects each in the matching placebo groups for these doses (10 subjects total received placebo).
Groups:
- PMN310 175 mg: PMN310 175 mg single IV infusion
- PMN310 350 mg: PMN310 350 mg single IV infusion
- PMN310 700 mg: PMN310 700 mg single IV infusion
- PMN310 1400 mg: PMN310 1400 mg single IV infusion
- PMN310 2800 mg: PMN310 2800 mg single IV infusion
- Placebo: Placebo
Period: Overall Study
Arm/Group | PMN310 175 mg | PMN310 350 mg | PMN310 700 mg | PMN310 1400 mg | PMN310 2800 mg | Placebo
Started | 6 | 6 | 6 | 6 | 6 | 10
Randomized Population | 6 | 6 | 6 | 6 | 6 | 10
Safety Population | 6 | 6 | 6 | 6 | 6 | 10
PK Population | 6 | 6 | 6 | 6 | 6 | 2
Evaluable Population | 6 | 6 | 6 | 6 | 6 | 10
Completed | 6 | 6 | 6 | 6 | 6 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PMN310 175 mg | PMN310 350 mg | PMN310 700 mg | PMN310 1400 mg | PMN310 2800 mg | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 6 | 6 | 10 | 40
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.50 (10.407) | 40.50 (9.854) | 46.17 (8.589) | 43.50 (8.826) | 41.67 (9.730) | 42.10 (10.671) | 42.08 (9.458)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 1 | 0 | 1 | 1 | 9
  Male | 4 | 2 | 5 | 6 | 5 | 9 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 5 | 0 | 2 | 6 | 24
  Not Hispanic or Latino | 0 | 1 | 1 | 6 | 4 | 4 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 6 | 4 | 1 | 14
  White | 5 | 4 | 5 | 0 | 2 | 9 | 25
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 6 | 6 | 6 | 10 | 40

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment Emergent Adverse Events
Description: Safety and tolerability of PMN310 following a single intravenous dose in healthy subjects.
Time Frame: 85 days
Measure: Number; unit: participants
Arm/Group | PMN310 175 mg | PMN310 350 mg | PMN310 700 mg | PMN310 1400 mg | PMN310 2800 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
participants
  Any TEAE | 2 | 2 | 0 | 3 | 3 | 3
  Any TEAE Related to Study Treatment | 1 | 1 | 0 | 0 | 1 | 2
  Any Severity Grade 3 TEAE | 1 | 0 | 0 | 0 | 1 | 1
  Any TESAE | 0 | 0 | 0 | 0 | 0 | 0
  Any TEAE Leading to Treatment Discontinuation | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Incidence of Clinically Significant Abnormal Findings in Laboratory Assessments (Hematology, Serum Clinical Chemistry, and Urinalysis)
Description: Safety and tolerability of PMN310 following a single intravenous dose in healthy subjects.
Time Frame: 85 days
Measure: Number; unit: participants
Arm/Group | PMN310 175 mg | PMN310 350 mg | PMN310 700 mg | PMN310 1400 mg | PMN310 2800 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
participants | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Incidence of Clinically Significant Abnormal Findings in Physical Examinations Including Neurological Examinations
Description: Safety and tolerability of PMN310 following a single intravenous dose in healthy subjects.
Time Frame: 85 days
Measure: Number; unit: participants
Arm/Group | PMN310 175 mg | PMN310 350 mg | PMN310 700 mg | PMN310 1400 mg | PMN310 2800 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
participants | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Incidence of Clinically Significant Abnormal Findings in Vital Signs (Supine Blood Pressure (BP), Pulse, Respiratory Rate and Oral Body Temperature)
Description: Safety and tolerability of PMN310 following a single intravenous dose in healthy subjects.
Time Frame: 85 days
Measure: Number; unit: participants
Arm/Group | PMN310 175 mg | PMN310 350 mg | PMN310 700 mg | PMN310 1400 mg | PMN310 2800 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
participants | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Incidence of Clinically Significant Abnormal Findings in 12 Lead Electrocardiogram (ECG)
Description: Safety and tolerability of PMN310 following a single intravenous dose in healthy subjects.
Time Frame: 85 days
Measure: Number; unit: abnormal findings
Arm/Group | PMN310 175 mg | PMN310 350 mg | PMN310 700 mg | PMN310 1400 mg | PMN310 2800 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
abnormal findings | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Summary of Serum Pharmacokinetic Parameters of PMN310 - AUCinf
Description: Measure concentration of PMN310 in serum
Time Frame: 0 to 2040 hours post-dose
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | PMN310 175 mg | PMN310 350 mg | PMN310 700 mg | PMN310 1400 mg | PMN310 2800 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
h*ng/mL | 19500000 (2680000) | 54800000 (24700000) | 91400000 (17200000) | 17300000 (26100000) | 417000000 (78400000)

7. Secondary Outcome: Summary of CSF Concentrations of PMN310
Description: Measure concentration of PMN310 in CSF
Time Frame: Days 3 and 29
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PMN310 175 mg | PMN310 350 mg | PMN310 700 mg | PMN310 1400 mg | PMN310 2800 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
ng/mL
  Day 3 | 50.05 (21.205) | 78.47 (35.281) | 150.10 (50.301) | 284.00 (136.995) | 502.50 (242.214)
  Day 29 | 32.43 (27.276) | 37.20 (19.916) | 92.80 (45.787) | 134.43 (71.353) | 241.00 (111.366)

8. Secondary Outcome: Summary of Serum Pharmacokinetic Parameters of PMN310 - AUClast
Description: Measure concentration of PMN310 in serum
Time Frame: 0 to 2040 hours post-dose
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | PMN310 175 mg | PMN310 350 mg | PMN310 700 mg | PMN310 1400 mg | PMN310 2800 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
h*ng/mL | 18900000 (2790000) | 49800000 (19600000) | 86300000 (16100000) | 16700000 (2440000) | 40000000 (71800000)

9. Secondary Outcome: Summary of Serum Pharmacokinetic Parameters of PMN310 - CL
Description: Measure concentration of PMN310 in serum
Time Frame: 0 to 2040 hours post-dose
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | PMN310 175 mg | PMN310 350 mg | PMN310 700 mg | PMN310 1400 mg | PMN310 2800 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
L/h | 0.00911 (0.00112) | 0.00737 (0.00281) | 0.00788 (0.00141) | 0.00824 (0.00134) | 0.00693 (0.00139)

10. Secondary Outcome: Summary of Serum Pharmacokinetic Parameters of PMN310 - Cmax
Description: Measure concentration of PMN310 in serum
Time Frame: 0 to 2040 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PMN310 175 mg | PMN310 350 mg | PMN310 700 mg | PMN310 1400 mg | PMN310 2800 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
ng/mL | 88300 (12800) | 350000 (171000) | 337000 (43600) | 704000 (33800) | 1480000 (201000)

11. Secondary Outcome: Summary of Serum Pharmacokinetic Parameters of PMN310 - T1/2
Description: Measure concentration of PMN310 in serum
Time Frame: 0 to 2040 hours post-dose
Measure: Mean (Standard Deviation); unit: h
Arm/Group | PMN310 175 mg | PMN310 350 mg | PMN310 700 mg | PMN310 1400 mg | PMN310 2800 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
h | 385.44 (52.07) | 491.61 (102.93) | 456.26 (61.45) | 440.09 (44.06) | 394.02 (111.30)

12. Secondary Outcome: Summary of Serum Pharmacokinetic Parameters of PMN310 - Tmax
Description: Measure concentration of PMN310 in serum
Time Frame: 0 to 2040 hours post-dose
Measure: Median (Full Range); unit: h
Arm/Group | PMN310 175 mg | PMN310 350 mg | PMN310 700 mg | PMN310 1400 mg | PMN310 2800 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
h | 2.25 [1.28 to 3.25] | 5.75 [1.75 to 37.42] | 1.75 [1.27 to 3.25] | 2.75 [1.35 to 37.25] | 7.25 [1.35 to 96.93]

13. Secondary Outcome: Summary of Serum Pharmacokinetic Parameters of PMN310 - Vd
Description: Measure concentration of PMN310 in serum
Time Frame: 0 to 2040 hours post-dose
Measure: Mean (Standard Deviation); unit: L
Arm/Group | PMN310 175 mg | PMN310 350 mg | PMN310 700 mg | PMN310 1400 mg | PMN310 2800 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
L | 5.08 (1.08) | 5.08 (1.96) | 5.22 (0.735) | 5.17 (0.419) | 4.32 (0.805)

14. Other Pre Specified Outcome: Immunogenicity of PMN310 - Anti-drug Antibodies (ADAs) in Serum
Description: The number of subjects who developed detectable levels of anti-PMN310 antibodies following a single intravenous dose
Time Frame: 85 days
Population: The number of subjects who developed detectable levels of anti-PMN310 antibodies following a single intravenous dose. Only subjects that were not confirmed ADA positive at Baseline were included in the overall tabulation.
Measure: Number; unit: participants
Arm/Group | PMN310 175 mg | PMN310 350 mg | PMN310 700 mg | PMN310 1400 mg | PMN310 2800 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
participants
  Day 85 - Screening Assay, Positive | 1 | 3 | 2 | 0 | 1 | 3
  Day 85 - Screening Assay, Negative | 5 | 3 | 4 | 6 | 5 | 7
  Day 85 - Confirmatory Assay, Positive | 0 | 3 | 0 | 0 | 1 | 1
  Day 85 - Confirmatory Assay, Negative | 1 | 0 | 2 | 0 | 0 | 2
  Overall - ADAs, Positive | 0 | 2 | 0 | 0 | 1 | 0
  Overall -ADAs, Negative | 5 | 3 | 6 | 6 | 5 | 9

ADVERSE EVENTS:
Time Frame: 85 days
Arm/Group | PMN310 175 mg | PMN310 350 mg | PMN310 700 mg | PMN310 1400 mg | PMN310 2800 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10
Other Adverse Events (participants affected / at risk) | 2/6 | 2/6 | 0/6 | 3/6 | 3/6 | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PMN310 175 mg (N=6) | PMN310 350 mg (N=6) | PMN310 700 mg (N=6) | PMN310 1400 mg (N=6) | PMN310 2800 mg (N=6) | Placebo (N=10)
Presyncope (Nervous system disorders) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute stress disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Application site hypersensitivity (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fracture treatment (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-09-22): https://cdn.clinicaltrials.gov/large-docs/28/NCT06105528/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-07): https://cdn.clinicaltrials.gov/large-docs/28/NCT06105528/SAP_001.pdf